CLINICAL TRIAL: NCT03999606
Title: Short-Term Music Training and Auditory Processing in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Assal Habibi, Assistant Research Professor of Psychology, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UP-19-00350
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Music Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Active Comparator): Participants in the control group will be assigned to a online based mindfulness training.
  Interventions: Behavioral: Music Training - Choir participation
- Music Training (Experimental): Participants in the experimental group will be assigned to a online based choir program.
  Interventions: Behavioral: Music Training - Choir participation

INTERVENTIONS:
Behavioral: Music Training - Choir participation — Sixty participants, ages 50-65, will be recruited to partake in this study and will be randomly assigned to two groups:
  participants in the experimental group will join a weekly on-line choir via Zoom, for ten weeks, directed by a professionally trained conductor from USC Department of Choral Music. The group practice will be accompanied by individual singing lessons (online or CDs) for home practice. Participants in the control group will be provided with weekly remote mindfulness lessons also on an online platform.

SUMMARY:
Most adults experience some degree of hearing loss by age 60. Hearing aids can improve some aspects of peripheral hearing but the loss of the ability to clearly perceive speech in noisy environments remains to be a significant deficit and often reduces life quality in older adults. Long-term music training has been shown to enhance auditory processing and specifically benefit speech-in-noise perception. It is not clear however whether short-term participation in a musically engaged activity can benefit such abilities in older adults. The proposed study aims to investigate whether short-term participation in a weekly community choir can improve speech in noise perception and its neural substrates as measured by sensory auditory evoked potentials (ERPs) to speech stimuli in older adults with mild to moderate subjective hearing loss. Sixty participants, ages 50-65, will be recruited to partake in this study and will be randomly assigned to two groups: participants in the experimental group will join a weekly remote choir on an on-line platform (Zoom), for ten weeks, directed by a professionally trained conductor from USC Department of Choral Music. The group practice will be accompanied by individual singing lessons (online or CDs) for home practice. Participants in the control group will be provided with weekly remote mindfulness lessons also on an on-line platform. All participants will be assessed remotely pre and post intervention, with behavioral measures of speech in noise perception and probes assessing emotional well-being and life satisfaction. Changes in auditory measures and their neural correlates and overall quality of life will be compared between the groups. The findings from this study can provide preliminary data to support a larger study on the impact of music engagement in improving the lives of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Native English speaker with experience of subjective hearing loss;
* Normal IQs (standard score of >85) as measured by the two-subtest Abbreviated Wechsler's Adult Scale of Intelligence.

Exclusion Criteria:

* Use of prescribed hearing aids;
* Sever hearing loss (thresholds of 60 and 95 dB)
* Current diagnosis of neurological or psychiatric disorders
* Impaired cognitive function (all participants will be screened with the Montreal Cognitive Assessment Battery)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 61 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Enhanced speech in noise perception | 15 weeks
  The effects of age on participants' ability to detect speech in noise will be assessed using the QuickSIN test (Speech-In-Noise; Version 1.3).
Enhanced speech in noise perception | 15 weeks
  EEG data will be collected using the speech syllable /da/, spoken in isolation by an American female. The stimulus will be presented in four conditions, in quiet and in presence of an 8-talker babble noise at three SNRs (10, 5 and 0 dB), presented in a random order for each participant, with an inter-stimulus interval of 1000 ms.

SECONDARY OUTCOMES:
Psychological Well-Being | 15 weeks
  Ryff's Psychological Well-Being Scale (2007) will be used to measure six aspects of wellbeing and happiness including autonomy, environmental mastery, personal growth, positive relations, purpose in life, and self-acceptance

CONTACTS AND LOCATIONS:
Locations (1):
- Brain and Creativity Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No